CLINICAL TRIAL: NCT05858619
Title: Molecular Signatures of Cutaneous Dupilumab Response
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-35748
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- dupilumab treatment (Experimental): Treatment with IL4RA inhibitor
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — dupilumab 600 mg injection initially and then 300 mg every other week

SUMMARY:
This study examines the effect of IL4RA blockade with dupilumab on the immune cells of atopic dermatitis skin lesions.

DETAILED DESCRIPTION:
This is a one-arm, open-label study to examine the effect of dupilumab. Dupilumab is a FDA-approved medication for the treatment of atopic dermatitis. This study will examine how dupilumab affects immune cells within atopic dermatitis skin lesions. Fifteen subjects with moderate to severe atopic dermatitis will be enrolled. Biopsy samples will be collected and undergo molecular profiling to correlate profiles with and to predict dupilumab treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. atopic dermatitis with a EASI (Eczema Area and Severity Index (EASI)) score of ≥7

Exclusion Criteria:

1. Known pregnancy
2. Known immunodeficiencies
3. Known parasitic infection -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Eczema Area and Severity Index (EASI) score from baseline to 8-12 weeks | baseline and 8-12 weeks
  Change in EASI score from baseline to 8-12 weeks. Scores range from 0 to 72, with higher scores indicating more severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cheng, MD, PhD, Principal Investigator — University of California, San Francisco; Raymond Cho, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No